CLINICAL TRIAL: NCT06798220
Title: Acute Effects of Ultra-processed Foods on Appetite Regulation in Individuals with Different Body Mass Indexes
Brief Title: Ultra-Processed Foods and Appetite Regulation: Acute Effects Across Body Mass Index Categories
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Menşure Nur ÇELİK, Principal Investigator, Ondokuz Mayıs University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B.30.2.ODM.0.20.08/663; 5085 (Other Grant/Funding Number: On Dokuz Mayıs University Scientific Research Project)
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Healthy Adult Volunteers
Keywords: ultra-processed foods; obesity; appetite regulation; incretins
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trad-breakfast (Experimental): Participants were served a traditional breakfast on the first experimental day.
  Interventions: Other: Traditional Breakfast
- UPF-breakfast (Experimental): Participants were served a ultra-processed breakfast on the second experimental day.
  Interventions: Other: UPF Breakfast

INTERVENTIONS:
Other: Traditional Breakfast — In this intervention, participants are offered a traditional breakfast (consisting of unprocessed or minimally processed foods), and postprandial appetite regulation is evaluated. Traditional breakfast includes chicken egg (boiled), white cheese (full-fat), white bread, black and green olives, tomatoes, cucumbers, and freshly squeezed orange juice.
  Arms: Trad-breakfast
Other: UPF Breakfast — In this intervention, participants are offered an ultra-processed breakfast, and postprandial appetite regulation is evaluated. Ultra-processed breakfast includes pan-fried beef sausage (without oil), packaged sandwich bread, tomato-based ketchup, and packaged orange juice.
  Arms: UPF-breakfast

SUMMARY:
This study was planned to observe the acute effects of minimally processed and ultra-processed food (UPF) consumption on appetite in participants with normal body mass index (BMI) [BMI: 18.5-24.99 kg/m2] and overweight-obese (BMI > 25 kg/m2) according to the NOVA (not an abbreviation) classification and to compare the postprandial effects of minimally processed and UPF consumption on appetite in normal and overweight-obese individuals. The study was designed as a non-randomized controlled, crossover study. The main questions it aims to answer are:

* Does a breakfast consisting of UPF affect appetite regulation differently compared to a breakfast consisting of unprocessed or minimally processed foods?
* Do the effects of foods with different levels of processing on appetite regulation vary by BMI?

Researchers will evaluate the effects of a breakfast containing unprocessed or minimally processed foods and a breakfast containing ultra-processed foods, which are similar in terms of energy and macronutrients, on appetite regulation.

Participants will:

* 1st experiment day: come to the laboratory where the experiment will be conducted at 8:00 am on an empty stomach and consume a breakfast containing unprocessed or minimally processed foods (chicken egg (boiled), white cheese (full-fat), black and green olive, tomato, cucumber, white bread, orange juice (freshly squeezed).
* 2nd experiment (after 2 weeks wash-out from 1st experiment): come to the laboratory where the experiment will be conducted at 8:00 am on an empty stomach and consume a breakfast containing ultra-processed food (packaged sandwich bread, beef sausage (pan-fried without oil), tomato ketchup, packaged orange juice).

DETAILED DESCRIPTION:
The study was conducted on adult participants between May 2024 and July 2024. The sample size was determined through power analysis to achieve 80% statistical at a two-sided significance level of 0.05, determining that a minimum of 25 participants were required for inclusion in the study. At this point, a total of 28 participants from both sexes were included in the study (20 female and 8 male participants). Participants aged 19 to 64 years were included in the study. On the other hand, participants were excluded from the study if they were pregnant or breastfeeding, in the premenstrual or menstrual phase, had food allergies or intolerances, followed specific dietary therapies, smoked, consumed alcohol chronically, were using probiotics and/or prebiotics, had any acute or chronic diseases, and were taking medications such as hormone replacement therapy, anticoagulants, antidepressants, antidiabetics, antihypertensives, antihyperlipidemic, or proton pump inhibitors. Ethics committee approval suitable for the Declaration of Helsinki was received from Ondokuz Mayıs University Clinical Research Ethics Committee (Ethics committee no: B.30.2.ODM.0.20.08/663). Volunteers were interviewed face-to-face, and a signed written consent form was obtained from each participant.

In the beginning of the study, the anthropometric measurements of the participants were assessed. Within the score, body weight and height were measured, and body composition was analyzed. The height measurements were taken without shoes, with the participants standing in the Frankfurt horizontal plane position (where the eye triangle and the top of the tragus are aligned on the same line). The weight measurements were determined using an electronic scale sensitive to 0.1 kg (Tanita MC-980). Moreover, the BMI (kg/m2) was calculated from body weight and height measurements. Participants were categorized based on their body mass index (BMI) as follows: normal BMI (18.5-24.99 kg/m2, n = 18) and high BMI (>25 kg/m2, n = 10). Waist circumference was measured using a non-flexible measuring tape at the midpoint between the iliac crest and the lowest rib, while hip circumference was measured parallel to the ground at the widest point on the hip using an inflexible measuring tape.

The participants included in the study completed the study by coming to two visits between May 2024 and July 2024. In these visits, two different breakfasts (Turkish traditional and ultra-processed breakfast) were served to participants, and then the impacts of these different breakfasts on postprandial appetite regulation were evaluated.

To determine the participants' food consumption prior to the experiment, semiquantitative Food Frequency Questionaries (FFQ) were taken for the last 3 months. Daily food intake was determined by multiplying the amounts of food consumed by the coefficients corresponding to the frequency of consumption. Additionally, to standardize the participants' dietary intake prior to the experiment, they were instructed to maintain a similar diet on the prior day of each visit. To verify compliance, 24-hour recall food consumption records were obtained from the participants for the day before both experimental days. The obtained data both from FFQ and 24-hour dietary recall were entered into the BEBIS (8.0) (Nutrition Information System) program to assess the energy and macro- and micronutrient intake of the participants.

Participants were instructed to arrive at the laboratory at 8:00 a.m. on the first test day in a fasting state. On this first test day, participants were served a Turkish traditional breakfast consisting of unprocessed or minimally processed foods. On the second test day after the 15-day wash-out period, participants were served a breakfast meal containing ultra-processed foods (UPF Breakfast). The traditional breakfast includes a chicken egg (boiled), white cheese (full-fat), white bread, black and green olives, tomatoes, cucumbers, and freshly squeezed orange juice. On the other hand, the UPF breakfast includes pan-fried beef sausage (without oil), packaged sandwich bread, tomato-based ketchup, and packaged orange juice. Both breakfasts were similar in terms of energy and macronutrient composition.

Participants were requested to arrive at the study laboratory by 8 a.m. on the day of the experiment with at least 12 hours of fasting. Breakfasts containing foods with similar energy and macronutrient composition but different levels of processing were served to participants. Participants were instructed to consume the entire breakfast within a 15-minute period. A visual analog scale (VAS) was used to subjectively assess postprandial appetite regulation. In this context, participants were requested to fill out the VAS at the beginning of the breakfast (0 min) and at 30, 60, 90, and 120 minutes after breakfast. The VAS form, completed at each time point, comprises four questions: [1] "How hungry do you feel?" [2] "How full do you feel?" [3] "How strong is your desire to eat?" and [4] "How much do you think you could eat?". Participants were instructed to indicate their response by marking the appropriate point along a 100-mm line, which was intentionally left unnumbered to avoid influencing their answers. The participants' responses to the questions were quantified by measuring the marked point on the 100-mm line using a ruler. The area under the curve was calculated using the numerical values obtained for each of the 4 questions at each time point from VAS.

To objectively evaluate postprandial appetite regulation, blood samples were collected at baseline (0 min) while participants were in a fasted state, as well as at 30, 60, 90, and 120 minutes following the first bite of breakfast. Serum was separated from whole blood, snap-frozen, and stored at -80°C until biochemical analysis. Within the scope, the levels of serum glucose were analyzed using glucose oxidase methods. Moreover, the serum levels of insulin, ghrelin, GLP1, GIP, and amylin (islet amyloid polypeptide) levels were quantified using a commercially available enzyme-linked immunosorbent assay (ELISA) kit (BT Lab, Shanghai, China). Using the analysis results obtained from biochemical analysis at each time point, the total AUC (tAUC) and incremental AUC (iAUC) values were calculated for the respective parameter.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.50-24.99 kg/m2 or > 25.00 kg/m2
* Not in premenstrual (1 week before menstruation) period or menstrual period for women participants

Exclusion Criteria:

* Being pregnant, breastfeeding, or postmenopausal
* Being in the premenstrual or menstruation phase
* Undergoing hormone replacement therapy
* Having an acute or chronic illness
* Taking regular medication (such as hormone replacement therapy, anticoagulants, antidepressants, antidiabetics, antihypertensives, antihyperlipidemics, proton pump inhibitors, etc.)
* Having a genetic and/or systemic disease
* Having any food allergies or intolerances
* Following a specific dietary regimen
* Smoking
* Consuming alcohol
* Having used antibiotics in the last 3 months
* Using prebiotics or probiotics
* Not giving consent after reading the informed consent form

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Changes in appetite-related hormones | At both the traditional breakfast and ultra-processed breakfast, blood samples were collected at the start of the both breakfasts and subsequently at the 30th, 60th, 90th, and 120th minutes.
  Evaluate the levels of fasting and postprandial changes by taking samples at regular intervals for two hours (at the start of both breakfasts and subsequently at the 30th, 60th, 90th, and 120th minutes) in appetite regulatory hormones such as insulin, ghrelin, glucagon-like peptid-1, gastric inhibitory peptide, and amylin (nM) through commercially available enzyme-linked immunosorbent assay (ELISA) kits.
Changes in visual analogue scale score | At both the traditional breakfast and ultra-processed breakfast, visual analogue scale was filled at the start of the both breakfasts and subsequently at the 30th, 60th, 90th, and 120th minutes.
  A visual analog scale (VAS) was used to subjectively assess postprandial appetite regulation. The VAS form, completed at each time point, comprises four questions: [1] "How hungry do you feel?" [2] "How full do you feel?" [3] "How strong is your desire to eat?" and [4] "How much do you think you could eat?". Participants were instructed to indicate their response by marking the appropriate point along a 100-mm line, which was intentionally left unnumbered to avoid influencing their answers. The participants' responses to the questions were quantified by measuring the marked point on the 100-mm line using a ruler.

SECONDARY OUTCOMES:
Changes in the energy received during the rest of the experimental day | After every two breakfasts for the rest of the day, one day for every two experimental days
  Participants were asked to record their food consumption for the rest of the day for both experimental days and the amount of energy they consumed (kcal) was calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University Kurupelit Campus, 55139 Atakum / SAMSUN, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided